CLINICAL TRIAL: NCT02309385
Title: A Randomized, Parallel Group, Double-masked, Active-controlled Phase 1/2 Clinical Trial to Evaluate the Efficacy and Safety of Dexamethasone Sodium Phosphate Visulex System for the Treatment of Non-infectious Anterior Uveitis
Brief Title: Safety and Efficacy Study of DSP-Visulex for the Treatment of Anterior Uveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aciont Inc (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSPV-201; R44EY014772 (NIH)
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Non-Infectious Anterior Uveitis
Keywords: uveitis; acute uveitis; anterior uveitis; dexamethasone sodium phosphate; non-infectious uveitis; DSP-Visulex; Aciont
MeSH Terms: conditions — Uveitis; Uveitis, Anterior | interventions — prednisolone acetate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 8% DSP-Visulex (Experimental): 8% dexamethasone sodium phosphate - Visulex (DSP- Visulex) and placebo eye drops in the affected eye.
  Interventions: Drug: 8% Dexamethasone Sodium Phosphate - Visulex
- 15% DSP-Visulex (Experimental): 15% dexamethasone sodium phosphate - Visulex (DSP- Visulex) and placebo eye drops in the affected eye.
  Interventions: Drug: 15% Dexamethasone Sodium Phosphate - Visulex
- Pred Forte (Active Comparator): Prednisolone acetate (1%) eye drops and vehicle - Visulex in the affected eye.
  Interventions: Drug: Prednisolone Acetate (1%) Eye Drops

INTERVENTIONS:
Drug: 8% Dexamethasone Sodium Phosphate - Visulex
  Other Names: 8% DSP- Visulex
  Arms: 8% DSP-Visulex
Drug: 15% Dexamethasone Sodium Phosphate - Visulex
  Other Names: 8% DSP- Visulex
  Arms: 15% DSP-Visulex
Drug: Prednisolone Acetate (1%) Eye Drops
  Other Names: Pred Forte
  Arms: Pred Forte

SUMMARY:
The purpose of this study is to determine the efficacy, safety, and tolerability of dexamethasone sodium phosphate Visulex (DSP-Visulex) after repeated-dose administration in patients with acute anterior uveitis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel group, double-masked, active- controlled study. Subjects will be enrolled and randomized to either 8 % or 15% DSP-Visulex with placebo drops or Vehicle-Visulex (V-Visulex) with prednisolone acetate 1% eye drops. All subjects will receive concomitant treatment with cyclopentolate.

ELIGIBILITY:
Inclusion Criteria:

* Non-infectious anterior uveitis

Exclusion Criteria:

* lntraocular pressure > 25mm Hg OU.
* Previous occurrence of an acute episode of anterior uveitis in affected eye(s) within 4 weeks prior to Visit 1.
* Historical or active intermediate or posterior uveitis in affected eye(s).
* Clear systemic causes of uveitis that may require or have required systemic treatment
* Uveitis suspected to have resulted from recent surgery or trauma.
* Use of ocular medication of any kind in affected eye(s) more than 2 days prior to Visit 1, excluding artificial tears, topical allergy medications, eyelid scrubs.
* Current use, or anticipated initiation during the study, of a corticosteroid or an immunosuppressant agent by any route (oral, inhaled, ocular, dermal). Current stable use is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with anterior chamber cell ACC grade of zero | Day 15

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events | 29 days
Proportion of patients with no uveitis symptoms | 29 days
Proportion of patients with improvement in visual acuity | 29 days
  Change in ETDRS letter score
Change from baseline in anterior chamber cell (ACC) grade | Day 8
Change from baseline in anterior chamber cell (ACC) grade | Day 15
Change from baseline in anterior chamber cell (ACC) grade | Day 29
Proportion of patients with anterior chamber cell ACC grade of zero | Day 8
Proportion of patients with anterior chamber cell ACC grade of zero | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: William I Higuchi, PhD, Principal Investigator — Aciont Inc
Locations (6):
- United States (6):
  - Massachusetts Eye Research and Surgery Institution (MERSI), Cambridge, Massachusetts
  - Charlotte Eye, Ear, Nose, and Throat Associates, Charlotte, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - B-Berger and Associates, Austin, Texas
  - Retina and Uveitis Consultants of Texas, San Antonio, Texas
  - Moran Eye Center, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang-Lin JE, Attar M, Acheampong AA, Robinson MR, Whitcup SM, Kuppermann BD, Welty D. Pharmacokinetics and pharmacodynamics of a sustained-release dexamethasone intravitreal implant. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):80-6. doi: 10.1167/iovs.10-5285. PMID 20702826
- [Background] Czock D, Keller F, Rasche FM, Haussler U. Pharmacokinetics and pharmacodynamics of systemically administered glucocorticoids. Clin Pharmacokinet. 2005;44(1):61-98. doi: 10.2165/00003088-200544010-00003. PMID 15634032
- [Background] Cunningham ET Jr, Wender JD. Practical approach to the use of corticosteroids in patients with uveitis. Can J Ophthalmol. 2010 Aug;45(4):352-8. doi: 10.3129/i10-081. PMID 20648092
- [Background] Gan IM, Ugahary LC, van Dissel JT, Feron E, Peperkamp E, Veckeneer M, Mulder PG, Platenkamp GJ, van Meurs JC. Intravitreal dexamethasone as adjuvant in the treatment of postoperative endophthalmitis: a prospective randomized trial. Graefes Arch Clin Exp Ophthalmol. 2005 Dec;243(12):1200-5. doi: 10.1007/s00417-005-0133-1. Epub 2005 Oct 19. PMID 16235062
- [Background] GORDON DM. Use of dexamethasone in eye disease. J Am Med Assoc. 1960 Jan 23;172:311-2. doi: 10.1001/jama.1960.03020040009003. No abstract available. PMID 13851186
- [Background] Miller DJ, Li SK, Tuitupou AL, Kochambilli RP, Papangkorn K, Mix DC Jr, Higuchi WI, Higuchi JW. Passive and oxymetazoline-enhanced delivery with a lens device: pharmacokinetics and efficacy studies with rabbits. J Ocul Pharmacol Ther. 2008 Aug;24(4):385-91. doi: 10.1089/jop.2007.0116. PMID 18665810
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Rohdewald P, Mollmann H, Barth J, Rehder J, Derendorf H. Pharmacokinetics of dexamethasone and its phosphate ester. Biopharm Drug Dispos. 1987 May-Jun;8(3):205-12. doi: 10.1002/bdd.2510080302. PMID 3593899
- [Background] Weijtens O, Feron EJ, Schoemaker RC, Cohen AF, Lentjes EG, Romijn FP, van Meurs JC. High concentration of dexamethasone in aqueous and vitreous after subconjunctival injection. Am J Ophthalmol. 1999 Aug;128(2):192-7. doi: 10.1016/s0002-9394(99)00129-4. PMID 10458175
- [Background] Weijtens O, Schoemaker RC, Cohen AF, Romijn FP, Lentjes EG, van Rooij J, van Meurs JC. Dexamethasone concentration in vitreous and serum after oral administration. Am J Ophthalmol. 1998 May;125(5):673-9. doi: 10.1016/s0002-9394(98)00003-8. PMID 9625551
- [Background] Weijtens O, Schoemaker RC, Romijn FP, Cohen AF, Lentjes EG, van Meurs JC. Intraocular penetration and systemic absorption after topical application of dexamethasone disodium phosphate. Ophthalmology. 2002 Oct;109(10):1887-91. doi: 10.1016/s0161-6420(02)01176-4. PMID 12359610
- [Background] Weijtens O, van der Sluijs FA, Schoemaker RC, Lentjes EG, Cohen AF, Romijn FP, van Meurs JC. Peribulbar corticosteroid injection: vitreal and serum concentrations after dexamethasone disodium phosphate injection. Am J Ophthalmol. 1997 Mar;123(3):358-63. doi: 10.1016/s0002-9394(14)70131-x. PMID 9063245